CLINICAL TRIAL: NCT01753258
Title: Outcomes of Delivery in Patients With Dyspareunia- A Prospective Study
Brief Title: Outcomes of Delivery in Patients With Dyspareunia
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Delivery-Dyspareunia-HMO-CTIL
Record Dates: First submitted 2012-12-12; First posted 2012-12-20 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Dyspareunia; Pregnancy; Provoked Vestibulodynia; Pelvic Floor Dysfunction
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Definite diagnosis of dyspareunia: Patients who report dyspareunia, and whose dyspareunia was evaluated prior to delivery by a caregiver experienced with sexual pain disorders, with definite diagnosis.
- No definite diagnosis of dyspareunia: Patients who report dyspareunia but were not evaluated prior to delivery or were evaluated inappropriately (i.e. "yeast infection" without cultures, "inflammation" and other vague definitions).
- Patients without dyspareunia: Patients without dyspareunia- those who report non painful sexual intercourse. This group of patients will be used as a control group.

SUMMARY:
The focus of this pilot study is to determine if a woman who experiences pain during sexual intercourse has a higher risk of complications during labor and delivery secondary to pelvic floor dysfunction, anxiety and intolerance towards pelvic examinations. Furthermore, it is unclear whether women with prepartum dyspareunia experience an improvement following vaginal delivery. While physicians may expect that vaginal birth improves dyspareunia due to the stretching effect on pelvic floor, to date, there is insufficient evidence to support this claim. The Investigators plan to prospectively study 200 patients at our Institution, collect information regarding birth and follow them, via questionnaires, regarding their dyspareunia postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. 200 nulliparous women admitted to the Labor and Delivery Department at the Hadassah Medical Center, above the age of 18.
2. Able and willing to read, understand, and sign the Informed Consent Form and questionnaire.
3. Agree to be contacted in the future to complete telephone questionnaires.

Exclusion Criteria:

1. Induction of labor
2. Placental abruption, placenta previa
3. Malpresentation
4. Non reassuring fetal heart rate upon admission
5. Any other contraindication for vaginal delivery
6. Multifetal pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous women admitted to the Labor and Delivery Department at the Hadassah Medical Center, above the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Obstetrical outcome of women with a history of dyspareunia | 3 months -1 year
  The Investigators will record the mode of delivery (vaginal, instrumental or cesarean section), length of the second stage of labor, use of anesthetics, perineal tears and\or episiotomies, and newborn's birth weight. The evaluation will be done prospectively, comparing data with matched controls without a history of dyspareunia.

SECONDARY OUTCOMES:
Rate of alleviation of dyspareunia following vaginal delivery as assessed through patient questionnaires. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel